CLINICAL TRIAL: NCT01569620
Title: Improving Colorectal Cancer (CRC) Screening for Diverse Hispanics in an Urban Primary Care Setting
Brief Title: Improving Colorectal Cancer Screening for Diverse Hispanics in Urban Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GCO 08-1159
Record Dates: First submitted 2012-03-29; First posted 2012-04-03 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Colorectal Cancer Screening
Keywords: Colorectal Cancer Screening; CRC; Screening Colonoscopy; Hispanics; Latinos

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Culturally targeted print materials (Active Comparator): Best clinical practices plus culturally print materials
  Interventions: Behavioral: Best clinical practices plus culturally targeted print materials
- Standard print materials (Active Comparator): Best clinical practices plus standard print materials
  Interventions: Behavioral: Best clinical practices plus standard print materials
- Best clinical practices alone (Active Comparator): Best clinical practices alone: This intervention arm includes best clinical practices (or standard/usual care at MSSM) and no additional print materials.
  Interventions: Behavioral: Best clinical practices alone

INTERVENTIONS:
Behavioral: Best clinical practices plus culturally targeted print materials — This intervention arm includes best clinical practices (or usual care at MSSM) and the culturally relevant print materials developed for this study.
  Arms: Culturally targeted print materials
Behavioral: Best clinical practices plus standard print materials — This intervention arm includes best clinical practices (or usual care at MSSM) and the standard CRC screening print materials developed by the Centers for Disease Control (CDC).
  Arms: Standard print materials
Behavioral: Best clinical practices alone — This intervention arm includes best clinical practices (or standard/usual care at MSSM) and no additional print materials.
  Other Names: Usual Care
  Arms: Best clinical practices alone

SUMMARY:
The proposed study seeks to investigate the impact of a culturally targeted print educational intervention on rates of colorectal cancer (CRC) screening via colonoscopy among Hispanics. If, as expected, the addition of culturally targeted materials to best clinical practices as compared to a) best clinical practices plus standard materials or b) best clinical practices alone leads to higher rates of CRC screening via colonoscopy then the culturally targeted print educational materials can be easily disseminated among this rapidly growing minority group who have low rates of CRC screening and whose disease is detected at later, less curable stages.

DETAILED DESCRIPTION:
CRC is the 2nd leading cause of cancer death among Hispanic women and men. Hispanics are more likely to be diagnosed at more advanced disease stages compared to non-Hispanic whites and have a lower probability of survival. A key way to decrease mortality from CRC among Hispanics is to increase rates of CRC screening and thereby early detection of CRC. To address low screening rates, thereby increasing the prevention and early detection of CRC, the proposed research seeks to increase CRC colonoscopy screening among Hispanics. The primary aim is to investigate the impact of a culturally targeted print educational intervention designed to increase CRC screening via colonoscopy in a diverse group of Hispanics 50 years of age and older. Our long standing (since 1999) research platform has included significant community input through ongoing meetings with our Community Advisory Board (CAB) soliciting their viewpoints and concerns. In addition, we consult with key community members on an ongoing basis for additional input. A Randomized Clinical Trial (RCT) will be conducted with 400 Hispanics within the context of the best clinical practices currently provided at Mount Sinai. There are three study arms: 1) best clinical practices plus culturally relevant print materials, 2) best clinical practices plus standard print materials and 3) best clinical practices alone. These three arms will allow the investigation of the addition of print materials and the comparison of culturally relevant to standard print materials to assess the differential impact of each print format. This comparison controls for the possible benefit of adding standard print materials to best clinical practices and allows for investigation of the additional benefit of culturally targeted relevant materials over and above that of standard materials. Further, by including feedback from the community, we will be able to clearly understand the benefits of, and be able to disseminate culturally targeted materials among this rapidly growing minority group. If, as hypothesized, the addition of the culturally targeted print materials leads to higher rates of colonoscopy, they can then be easily disseminated among health care settings treating Hispanics.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified Hispanic
* Between the ages of 50 and 85
* Able to provide informed consent in either English or Spanish
* No participation in study Focus Groups by a family member or oneself
* Referred for a screening colonoscopy by a primary care physician at Mount Sinai
* At average risk for developing colorectal cancer
* Have no colonoscopy procedure within the last 5 years
* Have telephone service

Exclusion Criteria:

* Personal history of CRC
* Personal history of any chronic GI disorder (irritable bowel syndrome, colitis) and
* Family history of CRC (first degree relative of CRC)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2012-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline of colonoscopy at 3 months, 6 months, and 12 months. | Baseline, at 3 months, at 6 months, and at 12 months
  Comparison of physician recommended colonoscopy (post intervention) obtained at approximately 3 months and 6 months (via self report) and at 12 months (as per chart review), to that of colonoscopy obtained at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine DuHamel, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Lina Jandorf, MA, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Cotter G, DuHamel K, Schofield E, Jandorf L. Processes of Change for Colonoscopy: Limited Support for Use Among Navigated Latinos. J Racial Ethn Health Disparities. 2019 Apr;6(2):327-334. doi: 10.1007/s40615-018-0528-4. Epub 2018 Oct 9. PMID 30302744